CLINICAL TRIAL: NCT07041684
Title: Microbiota and Lipedema: Weight Loss, Metabolic and Inflammatory Pattern, and Quality of Life in Obese Patients Before and After Treatment With Very Low Energy Ketogenic Vegan Therapy
Brief Title: Microbiota and Lipedema Evaluation in Obese Patient Treated With Very Low Energy Ketogenic Vegan Therapy
Acronym: MLVLEKVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Lucio Gnessi, Clinical Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLK24
Record Dates: First submitted 2024-12-15; First posted 2025-06-27 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2024-12

CONDITIONS: Lipedema; Obesity; Dysbiosis
MeSH Terms: conditions — Lipedema; Obesity; Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obese patients with lipedema (Experimental): Obese patients with lipedema treated with vegan VLEKT
  Interventions: Dietary Supplement: Very Low Energy Ketogenic Therapy with vegan meal replacements

INTERVENTIONS:
Dietary Supplement: Very Low Energy Ketogenic Therapy with vegan meal replacements — Metagenomics analysis of gut microbiota at baseline and after 45 days
  Other Names: Microbiota Analysis

SUMMARY:
Lipedema is a progressive, hereditary, multifactorial disease that occurs primarily in women, characterized by an abnormal and painful accumulation of subcutaneous fatty tissue. The etiology of lipedema is not entirely clear, but genetic, hormonal, vascular, and lymphatic factors have been implicated. Recent research suggests a potential role of the gut microbiota in the etiopathogenesis and progression of the disease, as alterations in gut microbial composition (dysbiosis) could contribute to chronic systemic inflammation and metabolic dysfunction that exacerbate the fat deposition typical of lipedema.

The condition is often associated with obesity, contributing to a state of chronic inflammation that exacerbates its progression. Among management strategies, Very Low Energy Ketogenic Therapy (VLEKT) has been proposed for its potential in improving inflammation and metabolism. VLEKT, an extremely low-calorie dietary regimen that induces ketosis through carbohydrate reduction, has been studied primarily for weight management, but the adoption of a plant-protein variant could offer additional benefits due to their anti-inflammatory properties resulting primarily from positive modulation of the gut microbiota.

The purpose of this study was to evaluate the effects of a plant protein-based ketogenic diet on the composition of the gut microbiota of obese patients with lipedema and to observe how it affected the symptoms of the condition. This experimental study analyzed anthropometric, metabolic, inflammatory parameters and the gut microbiota, as well as quality of life. The results obtained made it possible to evaluate the effectiveness of this dietary approach in the context of lipedema management, emphasizing the role of the gut microbiota and the anti-inflammatory properties of plant proteins. However, the single-center nature and limited number of participants represent limitations for generalizing the results.

Methods The present work is a prospective experimental study, in which a participant group consisting of 20 female individuals with lipedema were observed and offered plant protein-based VLEKT. Patients chosen to participate in the study were identified according to the following eligibility criteria: female subjects aged >18 years with a diagnosis of clinical stage II-III lipedema and with prior dietary treatment.

The presence of any of the following conditions prevented their enrollment in the study: subjects without an indication for treatment or unable to undergo VLEKT treatment; pregnancy and lactation; treatment with drugs interfering with proper microbiota analysis; and male subjects.

Each subject participating in the study underwent an initial outpatient specialist examination, and through the medical history, the following data were collected: age, sex, general and pathological health condition, and hematochemical parameters paying attention especially to CRP, blood glucose, insulin, total and HDL cholesterol, and triglycerides. Anthropometric parameters were then taken, including: weight; height; waist circumference; hip circumference; right and left thigh circumference; right and left arm circumference; right and left calf circumference; and right and left ankle circumference.

Once the anthropometric data were recorded, body composition analysis was conducted, which allowed the assessment of parameters such as: total water (TBW); extracellular water (ECW); intracellular water (ICW); lean body mass (FFM); and fat mass (FM).

Each patient received a fecal sample extraction kit in order to perform gut microbiota analysis. The same data were collected again at the end of the study after 45 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 30
* Female subjects aged > 18 years
* With a diagnosis of lipedema (II - III clinical stage)

Exclusion Criteria:

* Subjects without an indication for treatment
* Subjects who cannot undergo VLCKD treatment
* Pregnancy and lactation
* Treatment with drugs that interfere with proper microbiota analysis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2024-04-08 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
20 partecipants with changes in weight | From enrollment to the end of treatment at 45 days
  weight (kg)
20 partecipants with changes in BMI | From enrollment to the end of tratment at 45 days
  BMI - Body Mass Index (weight and height will be combined to report BMI in kg/m^2) whose ranges are: underweight (<18.5), normal weight (18.5-24.9), overweight (25-29.9), obesity (30 or more);
20 partecipants with changes in circumferences | From enrollment to the end of treatment at 45 days
  waist circumference (cm); hip circumference (cm); right and left thigh circumference (cm); right and left arm circumference (cm); right and left calf circumference (cm); and right and left ankle circumference (cm).
20 partecipants with changes in blood count | From enrollment to the end of treatment at 45 days
20 partecipants with changes in blood glucose, total and HDL cholesterol, and triglycerides | From enrollment to the end of treatment at 45 days
  blood glucose (mg/dL), total and HDL cholesterol (mg/dL), and triglycerides (mg/dL)
20 partecipants with changes in c-reactive protein (CPR) | From enrollment to the end of treatment at 45 days
  CPR (mg/L)
20 partecipants with changes in erythrocyte sedimentation rate (ESR) | From enrollment to the end of treatment at 45 days
  ESR (mm/h)
20 partecipants with changes in insulin | From enrollment to the end of treatment at 45 days
  insulin (µU/mL)
20 partecipants with changes in HOMA-INDEX | From enrollment to the end of treatment at 45 days
  HOMA-INDEX (threshold of 2.5)
20 partecipants with changes in body water (Total Body Water, Extracellular Water, Intracellular Water) by means of bioimpedance analysis (Akern BIVA 101) | From enrollment to the end of treatment at 45 days
  Total Body Water (L), Extracellular Water (L), Intracellular Water (L)
20 partecipants with changes in Free Fat Mass, Fat Mass, Body Cell Mass by means of bioimpedance analysis (Akern BIVA 101) | From enrollment to the end of treatment at 45 days
  Free Fat Mass (Kg), Fat Mass (Kg), Body Cell Mass (Kg)
20 partecipants with changes in Skeletal Muscle Index by means of bioimpedance analysis (Akern BIVA 101) | From enrollment to the end of treatment at 45 days
  Skeletal Muscle Index (>7,0 kg/m^2 in men and >5,7 kg/m^2 in women)
Short form of the McGill Pain Questionnaire (SF-MPQ) | From enrollment to the end of treatment at 45 days
  The main component of the SF-MPQ consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0 = none, 1 = mild, 2 = moderate or 3 = severe. Three pain scores are derived from the sum of the intensity rank values of the words chosen for sensory, affective and total descriptors. The SF-MPQ also includes the Present Pain Intensity (PPI) index of the standard MPQ and a visual analogue scale (VAS) from 0-100, where 100 is fort pain.
EuroQoL 5D (EQ-5D) | From enrollment to the end of treatment at 45 days
  The EQ-5D consists of five questions (also known as dimensions (5D): mobility, selfcare, usual activities, pain/discomfort, anxiety/depression) with 5 levels (5L) of problem severity in the responses, as well as a Visual Analogue Scale (EQ-VAS) aiming to capture a respondents' rating of their 'health today' on a scale from 0-100, where 100 is better health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Lucio Gnessi, Medical Doctor, Principal Investigator — University of Roma La Sapienza
Locations (1):
- La Sapienza, University of Rome, Rome, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basciani S, Camajani E, Contini S, Persichetti A, Risi R, Bertoldi L, Strigari L, Prossomariti G, Watanabe M, Mariani S, Lubrano C, Genco A, Spera G, Gnessi L. Very-Low-Calorie Ketogenic Diets With Whey, Vegetable, or Animal Protein in Patients With Obesity: A Randomized Pilot Study. J Clin Endocrinol Metab. 2020 Sep 1;105(9):dgaa336. doi: 10.1210/clinem/dgaa336. PMID 32484877
- [Background] Keith L, Seo CA, Rowsemitt C, Pfeffer M, Wahi M, Staggs M, Dudek J, Gower B, Carmody M. Ketogenic diet as a potential intervention for lipedema. Med Hypotheses. 2021 Jan;146:110435. doi: 10.1016/j.mehy.2020.110435. Epub 2020 Nov 27. PMID 33303304
- [Background] Caprio M, Infante M, Moriconi E, Armani A, Fabbri A, Mantovani G, Mariani S, Lubrano C, Poggiogalle E, Migliaccio S, Donini LM, Basciani S, Cignarelli A, Conte E, Ceccarini G, Bogazzi F, Cimino L, Condorelli RA, La Vignera S, Calogero AE, Gambineri A, Vignozzi L, Prodam F, Aimaretti G, Linsalata G, Buralli S, Monzani F, Aversa A, Vettor R, Santini F, Vitti P, Gnessi L, Pagotto U, Giorgino F, Colao A, Lenzi A; Cardiovascular Endocrinology Club of the Italian Society of Endocrinology. Very-low-calorie ketogenic diet (VLCKD) in the management of metabolic diseases: systematic review and consensus statement from the Italian Society of Endocrinology (SIE). J Endocrinol Invest. 2019 Nov;42(11):1365-1386. doi: 10.1007/s40618-019-01061-2. Epub 2019 May 20. PMID 31111407